CLINICAL TRIAL: NCT00857558
Title: A Phase 2 Study of OPC-262 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 262-08-001; JapicCTI-090697 (Other: JAPIC)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): OPC-262 1mg
  Interventions: Drug: saxagliptin
- 2 (Experimental): OPC-262 2.5mg
  Interventions: Drug: saxagliptin
- 3 (Experimental): OPC-262 5mg
  Interventions: Drug: saxagliptin
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: saxagliptin — orally administration at 1 mg once a day for 12 weeks
  Arms: 1
Drug: saxagliptin — orally administration at 2.5 mg once a day for 12 weeks
  Arms: 2
Drug: saxagliptin — orally administration at 5 mg once a day for 12 weeks
  Arms: 3
Drug: placebo — orally administration once a day for 12 weeks
  Arms: 4

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, group-comparison study to investigate the safety and efficacy of OPC-262 in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with HbA1c above 7.0% and below 10%
* Patients who are capable of giving informed consent
* Patients who are able to take contraceptive measures to avoid pregnancy of the patient or the patient's partner

Exclusion Criteria:

* Patients with type1 diabetes mellitus, patients with diabetes mellitus or impaired glucose tolerance (IGT) due to other specified mechanism or diseases, and patients with gestational diabetes mellitus
* Patients with a medical history of diabetes coma
* Patients with poorly-controlled hypertension
* Patients with heart failure
* Patients with a complication of active hepatitis or hepatic cirrhosis
* Patients undergoing treatment of glomeruler diseases other than diabetic nephropathy
* Patients with a history or complication of malignant tumor

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
changes in HbA1C from baseline | 2w, 4w, 8w, 12w, 16w

SECONDARY OUTCOMES:
values and changes in HbA1c form baseline | 2w, 4w, 8w, 12w, 16w
values and changes in fasting blood glucose (FSB) from baseline | 2w, 4w, 8w, 12w, 16w
adverse event | at any time

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — OPC-J
Locations (8):
- Japan (8):
  - Chubu Regin
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region